CLINICAL TRIAL: NCT04274062
Title: Effects of Peri Partum Integrated Nursing Care Versus Routine Care in Placenta Previa : A Randomized Controlled Trail
Status: Completed | Type: Observational
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Other Study IDs: Randomized controlled trial
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Placenta Previa Total; Nursing Role
Keywords: placenta previa; Nursing; antepartum hemorrhage; randomized trial
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- peri partum integrated nursing care of placenta previa: * Part (1) personal data:
  * Part (2) baseline and characteristics of the patients participants:
  * Tool II- An observation checklist: This tool is develop by researcher according to guideline of Royal College of Obstetricians and Gynaecologists, 2018), and divide into three main parts: preoperative, intraoperative and postoperative.
  * Part (1) pre-operative: includes assessment of :
  * patients general condition
  * investigation
  * reserved blood
  * Hemoglobin level
  * Impact of hysterectomy option. -9-
  Part (2) Intra-operative:
  Includes assessment of :-
  * Investigation
  * Vital signs
  * Hypothermia
  * Blood loss
  * I.V fluid
  * Blood gases
  * Fetal condition and APGAR score.
  * Part (3) Post-operative: Includes:
  * maternal complication
  * fetal complication
  * psychological satisfaction
  Interventions: Procedure: Integrated Nursing care of placenta previa
- peri partum regular care of placenta previa: Routine nursing care of all cases of placenta previa (preoperative, intraoperative and postoperative)..
  Interventions: Procedure: Integrated Nursing care of placenta previa

INTERVENTIONS:
Procedure: Integrated Nursing care of placenta previa — Phase I :( preparation phase) Phase II: (Implementation phase) includes Preoperative care , intraoperative care and postoperative care by a nurse.
  Phase III: (Evaluation phase)

SUMMARY:
At our institution, the annual number of placenta previa was 494 cases (1.7%); of whom 95 cases (19.2%) were proved to have a placenta accreta. Perioperatively, they are subjected to regular care of a tertiary university hospital. This study aims to determine the effectiveness of peri partum integrated nursing care for the patients with placenta previa versus routine care.

DETAILED DESCRIPTION:
Study design:

Experimental design: (randomized control trail)

Setting:

This study will be conducted at Woman's Health Hospital, Assiut University, emergency department and inpatient department.

Sample:

A convenience sample will be used, the total sample will include (100) patients with placenta previa, divided into two group1:1

* group 1: 50 patients study group
* group2: 50 patients control group

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with diagnosis of placenta previa.

Exclusion Criteria:

* Other high risk pregnancy cases

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant Placenta previa
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Improved maternal and fetal well beings in cases of placenta previa | 2 years
  Adding an integrated nursing care to the regular care of cases of placenta previa

CONTACTS AND LOCATIONS:
Overall Officials: Atef Darwish, Principal Investigator — Woman's Health University Hospital
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No